CLINICAL TRIAL: NCT04085146
Title: The Effect of Ventilation With Individualized Optimal Positive End Expiratory Pressure on Postoperative Atelectasis in Patients Undergoing Robot Assisted Laparoscopic Radical Prostatectomy
Brief Title: Individual Optimal Positive End-expiratory Pressure During Robot-assisted Laparoscopic Radical Prostatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Won Ho Kim, MD, Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1908-022-105
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Atelectasis, Postoperative
Keywords: robot-assisted surgery; prostatectomy; laparoscopy; positive end-expiratory pressure; individualized; atelectasis; general anesthesia
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Intervention Model Description: Randomized controlled superiority trial with two arms of intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Anesthesia care-provider cannot be blinded. Surgeon and outcome assessor will be blinded to the group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal PEEP (Experimental): Individualized optimal PEEP will be provided during the laparoscopic period of surgery. Optimal PEEP will be determined by the automated procedure of step-wised decrease in the amount of PEEP of the anesthesia ventilator Aisys Care Station (GE Healthcare, Madison, Wisconsin, USA).
  Interventions: Procedure: Individualized optimal positive end-expiratory pressure
- Conventional PEEP (Active Comparator): A same amount of PEEP of 7 centimeter hydrogen dioxide will be provided during the laparoscopic period of surgery.
  Interventions: Procedure: Conventional positive end-expiratory pressure

INTERVENTIONS:
Procedure: Individualized optimal positive end-expiratory pressure — Optimal PEEP will be determined by the automated procedure of step-wised decrease in the amount of PEEP of the anesthesia ventilator Aisys Care Station (GE Healthcare, Madison, Wisconsin, USA).
  Arms: Optimal PEEP
Procedure: Conventional positive end-expiratory pressure — A same amount of PEEP of 7 centimeter hydrogen dioxide will be provided during the laparoscopic period of surgery.
  Arms: Conventional PEEP

SUMMARY:
During robot-assisted radical prostatectomy, pneumoperitoneum with Trendelenburg position is used. However, perioperative atelectasis and respiratory complications may occur with high incidence due to general anesthesia and carbon dioxide pneumoperitoneum. Intraoperative ventilatory strategy to address these issues include intraoperative recruitment maneuver and positive end-expiratory pressure (PEEP). Recently, individualized optimal PEEP with minimal driving pressure or maximal respiratory compliance was reported to reduce respiratory complications after general anesthesia. A recent version of general anesthesia ventilator provides a stepwise procedure of determining optimal PEEP by calculating respiratory compliance. We investigated whether the application of individualized optimal PEEP could reduce the incidence of atelectasis and respiratory complications after robot-assisted laparoscopic radical prostatectomy compared to uniform PEEP.

DETAILED DESCRIPTION:
During robot-assisted radical prostatectomy, pneumoperitoneum with Trendelenburg position is used. However, perioperative atelectasis and respiratory complications may occur with high incidence due to general anesthesia and carbon dioxide pneumoperitoneum. Intraoperative ventilatory strategy to address these issues include intraoperative recruitment maneuver and positive end-expiratory pressure (PEEP). Recently, individualized optimal PEEP with minimal driving pressure or maximal respiratory compliance was reported to reduce respiratory complications after general anesthesia. A recent version of general anesthesia ventilator provides a stepwise procedure of determining optimal PEEP by calculating respiratory compliance. We investigated whether the application of individualized optimal PEEP could reduce the incidence of atelectasis and respiratory complications after robot-assisted laparoscopic radical prostatectomy compared to uniform PEEP. We plan to determine the degree of immediate postoperative atelectasis by measuring the lung ultrasound score and compare the lung ultrasound score between groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing robot-assisted laparoscopic radical prostatectomy
* Patients receiving mechanical ventilation by Aisys Care Station anesthesia ventilator
* Patients who provided written informed consent to participate in this clinical trial

Exclusion Criteria:

* American Society of Anesthesiologists physical status classification class 3 or more
* Moderate or more obstructive or restrictive pulmonary disease
* Preoperative adult respiratory distress syndrome or previous history of adult respiratory distress syndrome
* history of heart failure, unstable angina, increased intracranial pressure
* history of pneumothorax or presence of bullae

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2020-08-07 (Actual)

PRIMARY OUTCOMES:
Difference in lung ultrasound score | 10 min after surgery
  Difference in postoperative lung ultrasound score and baseline lung ultrasound score

SECONDARY OUTCOMES:
Baseline lung ultrasound score | 10 min before the start of anesthesia induction
  A scoring system with a sum of the B-line score and consolidation score by lung ultrasound examination
Composite of respiratory complication | during postoperative seven days.
  summation of the following events: hypoxemia (pulse oximetry of 95% or less), laryngospasm, bronchospasm, pneumonia, pulmonary infiltration, aspiration pneumonia, pneumonia), pulmonary infiltration, aspiration pneumonia, development of acute respiratory distress syndrome, atelectasis, pleural effusion, pulmonary edema, pneumothorax.
Length of hospital stay | during the postoperative one month
  Length of total hospital stay
Postoperative Lung ultrasound score | 10 min after the end of anesthesia
  A scoring system with a sum of the B-line score and consolidation score by lung ultrasound examination
Length of intensive care unit stay | during the postoperative one month
  Length of total hospital stay
Surgical wound infection | during the postoperative one month
  The rate of surgical wound infection
Surgical wound dehiscence | during the postoperative one month
  The rate of surgical wound dehiscence
Incidence of acute kidney injury | during the postoperative one month
  Incidence of postoperative acute kidney injury
Incidence of surgical re-intervention | during the postoperative one month
  Incidence of surgical re-open

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No